CLINICAL TRIAL: NCT01862471
Title: Improved Lower Limb Haemodynamics Using Neuromuscular Electrical Stimulation (NMES); Potential Novel DVT Prophylaxis
Brief Title: Neuromuscular Electrical Stimulation Versus Intermittent Pneumatic Compression for Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EE-NMES-DVT-012
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Venous Thrombosis
Keywords: Deep Vein Thrombosis; Neuromuscular Electrical Stimulation; Intermittent Pneumatic Compression; Doppler Ultrasound
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVT prophylaxis (Experimental): Neuromuscular electrical stimulation using a custom-built, two-channel stimulator (Duo-STIM (stimulator), Bioelectronics Research Cluster, National University of Ireland, Galway) with a frequency of 36 Hz, a balanced biphasic waveform with a pulse width of 350μs, a ramp up time of 500ms, a contraction time of 1s and a ramp down time of 500ms. Stimulation was applied every 20 seconds over a period of 5 minutes.
  Intermittent pneumatic compression using the Novamedix A-V Impulse System Model 6000 (Novamedix distribution Limited, England), programmed to deliver compression every 20 seconds at a pressure of 130 mmHg for a 1 second duration over a period of 5 minutes.
  Interventions: Device: Neuromuscular Electrical Stimulation; Device: Intermittent Pneumatic Compression

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Frequency of 36Hz, a balanced biphasic waveform with a pulse width of 350μs, a ramp up time of 500ms, a contraction time of 1s and a ramp down time of 500ms.
  Other Names: Custom-built, two-channel stimulator (Duo-STIM, Bioelectronics Research Cluster, NUI Galway)
Device: Intermittent Pneumatic Compression — Programmed to deliver compression every 20 seconds at a pressure of 130mmHg for a 1 second duration over a period of 5 minutes.
  Other Names: Novamedix AV Impulse System Model 6000 (Novamedix distribution Limited, England)

SUMMARY:
Deep Vein Thrombosis (DVT) is a life threatening condition and a serious concern among hospitalized patients, with death occurring in approximately 6% of cases. It involves the formation of a clot where stagnant blood flow occurs, predominantly in the deep veins of the legs. Three mechanisms underlie DVT, venous stasis (slowing or stopping of the blood), hypercoagulability (increased clotting) and damage to blood vessel endothelium (damage to blood vessel wall), collectively known as Virchow's triad.

Intermittent pneumatic compression (IPC) and neuromuscular electrical stimulation (NMES) have been shown to improve lower limb blood flow. However, few studies have directly compared the two methods and those that have, have used outdated NMES devices.

The objective of this study is to compare the effectiveness of a modern NMES device to intermittent pneumatic compression in terms of blood flow.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* History of heart/respiratory problems
* Pregnancy
* Presence of implants, including cardiac pacemakers and orthopaedic implants
* History of neurological disorder
* History of severe arterial disease or known dermatological problems
* Under 18 years of age or over 40 years of age

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Blood Flow Measurements from the Lower Limb | An hour and a half (plus or minus half an hour)

SECONDARY OUTCOMES:
Blood Pressure | An hour and a half (plus or minus half an hour)
Heart Rate | An hour and a half (plus or minus half an hour)

CONTACTS AND LOCATIONS:
Overall Officials: Gearoid OLaighin, PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- National University of Ireland, Galway, Galway, Ireland